CLINICAL TRIAL: NCT06127433
Title: The Effect of Short-term Insulin Intensive Therapy Based on the Application of Insulin Pump and Real-time Dynamic Glucose Monitoring Technology on Reversing the Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-816
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Insulin Pump，Continuous Glucose Monitoring Technology
MeSH Terms: interventions — Insulin Glargine; Metformin; dapagliflozin; Insulin Aspart

STUDY DESIGN:
Intervention Model Description: basal insulin and oral antidiabetic drugs group insulin intensive therapy group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Intervention：insulin pump intensive therapy
  Interventions: Drug: Insulin aspart
- control group (Active Comparator): basal insulin and oral antidiabetic drugs
  Interventions: Drug: Insulin Glargine; Drug: Metformin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Insulin Glargine — Insulin Glargine
  Arms: control group
Drug: Metformin — Metformin
  Arms: control group
Drug: Dapagliflozin — Dapagliflozin
  Arms: control group
Drug: Insulin aspart — Insulin aspart
  Arms: intervention group

SUMMARY:
This study aims to explore the effectiveness and safety of the in-hospital-out-of-hospital synergistic short-term insulin intensive therapy model based on patch insulin pump and continuous glucose monitoring technology through a randomized controlled study, and evaluate the possibility of blood glucose parameters derived from continuous glucose technology in predicting long-term blood glucose remission, so as to provide important reference data for the precision, intelligence, and integrated improvement of short-term insulin intensive therapy.

ELIGIBILITY:
Inclusion Criteria:1: Have never received any hypoglycemic treatment (including oral hypoglycemic drugs, traditional Chinese medicine hypoglycemic drugs, insulin) Type 2 diabetes patients, or type 2 diabetes patients with diagnosis time less than 1 year, use hypoglycemic drugs No more than 1 type, with a usage time of no more than 1 week, and discontinuation of medication for more than 1 week when selected

2: A1c of glycosylated hemoglobin ≥ 8.0%, and abdominal blood glucose>7.0mmol/L during enrollment

3: Age range from 18 to 70 years old, with a body mass index (BMI) of 20-35kg/m2

4: agrees to use contraception during the study process

5: Able and willing to use a dynamic blood glucose system and monitor blood glucose according to project requirements, and accept out of hospital lifestyle management and insulin hypoglycemic management.

-

Exclusion Criteria:1: Not type 2 diabetes

2: The medication used is allergic or intolerable

3: Acute complications of diabetes

4: Severe microvascular complications

5: Severe macrovascular complications

6: Blood pressure consistently exceeds 180/110mmHg and cannot be controlled within 160/110mmHg within 1 week

7: The clearance rate of blood creatinine is less than 45ml/min/1.73m2, the ALT is ≥ 3 times the normal upper limit, and the total bilirubin is ≥ 2 times the normal upper limit and lasts for more than 1 week

8: Hemoglobin<100g/L or requires regular blood transfusion treatment

9: Accumulated time of using drugs that may affect blood sugar within 12 weeks for more than 1 week

10: Systemic infection or severe accompanying diseases

11: Patients with malignant tumors or chronic diarrhea

12: Uncontrolled endocrine gland dysfunction

13: Mental disorders

14: Chronic heart failure, with a heart function grading of III or above

15: Pregnant, breastfeeding, women of childbearing age who are unwilling to use contraception during the study period, or have surgery plans that require general anesthesia in the near future (within 6 months)

16: The subject is uncooperative, unable to follow up, or the researcher determines that it may be difficult to complete the study.

17: Other situations that the researcher determines are not suitable for inclusion

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Intergroup remission rate at 24 week | 24 week
  Fasting blood glucose<7mmol/L, and glycated hemoglobin<6.5%

CONTACTS AND LOCATIONS:
Locations (1):
- 刘烈华, Guandong, China

IPD SHARING:
Plan to Share IPD: Yes